CLINICAL TRIAL: NCT02822599
Title: The Role of Human Fibrinogen Concentrate (RiaSTAP) in Decreasing Blood Loss and the Need for Component Blood Therapy in Infants Undergoing Cardiopulmonary Bypass.
Brief Title: Human Fibrinogen Concentrate in Pediatric Cardiac Surgery
Acronym: RiaSTAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicklaus Children's Hospital f/k/a Miami Children's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Tirotta, MD, MBA, Director Cardiac Anesthesia, Nicklaus Children's Hospital f/k/a Miami Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCH0000201496
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-06

CONDITIONS: Hypofibrinogenemia; Afibrinogenemia; Bleeding Disorders
Keywords: CBP, congenital heart defects, cardiopulmonary bypass
MeSH Terms: conditions — Afibrinogenemia; Hemostatic Disorders; Rubinstein-Taybi Syndrome; Heart Defects, Congenital | interventions — Fibrinogen; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RiaSTAP (Active Comparator): Group 1 will receive an infusion of RiaSTAP after termination of CPB at a dose of 70 mg/kg after randomization to this group.
  Interventions: Drug: RiaStAP
- Saline (Placebo Comparator): Group 2 will receive a placebo consisting of Normal Saline 0.9% (NS) after randomization to this group.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: RiaStAP — To decrease post-operative bleeding volume.
  Other Names: Fibrinogen Concentrate Human
  Arms: RiaSTAP
Drug: Saline — Placebo consisting of normal saline 0.9%
  Other Names: Normal Saline 0.9%
  Arms: Saline

SUMMARY:
The goal of the study is to determine whether the use of Human Fibrinogen Concentrate (RiaSTAP) will decrease blood loss and the need for component blood therapy in neonates and infants undergoing cardiopulmonary bypass.

DETAILED DESCRIPTION:
The goal of the study is to determine whether the use of Human Fibrinogen Concentrate (RiaSTAP) will decrease blood loss and the need for component blood therapy in neonates and infants undergoing cardiopulmonary bypass. RiaSTAP will be administered after termination of Cardiopulmonary Bypass (CPB) at a dose of 70 mg/kg, in a prospective, randomized, controlled study. We hypothesize that the administration of RiaSTAP in this manner will reduce peri-operative bleeding and transfusion requirements.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal and infant cardiac patients presenting for open-heart surgery at Nicklaus Children's Hospital will be eligible for enrollment in the study.

Exclusion Criteria:

* Patients who fall outside of the age range for the study will be excluded. Patients known to have had an anaphylactic or severe reaction to the drug or its components will not be enrolled. At the time of the rewarming ROTEM, any patient with a FIBTEM MCF > 15mm, will be excluded.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Tirotta, MD, Principal Investigator — Director Cardiac Anesthesia
Locations (2):
- United States (2):
  - Nickalus Children's Hospital f/k/a Miami Children's Hospital, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dacey LJ, Munoz JJ, Baribeau YR, Johnson ER, Lahey SJ, Leavitt BJ, Quinn RD, Nugent WC, Birkmeyer JD, O'Connor GT. Reexploration for hemorrhage following coronary artery bypass grafting: incidence and risk factors. Northern New England Cardiovascular Disease Study Group. Arch Surg. 1998 Apr;133(4):442-7. doi: 10.1001/archsurg.133.4.442. PMID 9565127
- [Background] Moulton MJ, Creswell LL, Mackey ME, Cox JL, Rosenbloom M. Reexploration for bleeding is a risk factor for adverse outcomes after cardiac operations. J Thorac Cardiovasc Surg. 1996 May;111(5):1037-46. doi: 10.1016/s0022-5223(96)70380-x. PMID 8622301
- [Background] Paparella D, Brister SJ, Buchanan MR. Coagulation disorders of cardiopulmonary bypass: a review. Intensive Care Med. 2004 Oct;30(10):1873-81. doi: 10.1007/s00134-004-2388-0. Epub 2004 Jul 24. PMID 15278267
- [Background] Miller BE, Tosone SR, Guzzetta NA, Miller JL, Brosius KK. Fibrinogen in children undergoing cardiac surgery: is it effective? Anesth Analg. 2004 Nov;99(5):1341-1346. doi: 10.1213/01.ANE.0000134811.27812.F0. PMID 15502028
- [Background] Kern FH, Morana NJ, Sears JJ, Hickey PR. Coagulation defects in neonates during cardiopulmonary bypass. Ann Thorac Surg. 1992 Sep;54(3):541-6. doi: 10.1016/0003-4975(92)90451-9. PMID 1510523
- [Background] Chan AK, Leaker M, Burrows FA, Williams WG, Gruenwald CE, Whyte L, Adams M, Brooker LA, Adams H, Mitchell L, Andrew M. Coagulation and fibrinolytic profile of paediatric patients undergoing cardiopulmonary bypass. Thromb Haemost. 1997 Feb;77(2):270-7. PMID 9157580
- [Background] Karlsson M, Ternstrom L, Hyllner M, Baghaei F, Nilsson S, Jeppsson A. Plasma fibrinogen level, bleeding, and transfusion after on-pump coronary artery bypass grafting surgery: a prospective observational study. Transfusion. 2008 Oct;48(10):2152-8. doi: 10.1111/j.1537-2995.2008.01827.x. Epub 2008 Jul 24. PMID 18657083
- [Background] Karlsson M, Ternstrom L, Hyllner M, Baghaei F, Flinck A, Skrtic S, Jeppsson A. Prophylactic fibrinogen infusion reduces bleeding after coronary artery bypass surgery. A prospective randomised pilot study. Thromb Haemost. 2009 Jul;102(1):137-44. doi: 10.1160/TH08-09-0587. PMID 19572078
- [Background] Rahe-Meyer N, Pichlmaier M, Haverich A, Solomon C, Winterhalter M, Piepenbrock S, Tanaka KA. Bleeding management with fibrinogen concentrate targeting a high-normal plasma fibrinogen level: a pilot study. Br J Anaesth. 2009 Jun;102(6):785-92. doi: 10.1093/bja/aep089. Epub 2009 May 2. PMID 19411671
- [Derived] Tirotta CF, Lagueruela RG, Gupta A, Salyakina D, Aguero D, Ojito J, Kubes K, Hannan R, Burke RP. A Randomized Pilot Trial Assessing the Role of Human Fibrinogen Concentrate in Decreasing Cryoprecipitate Use and Blood Loss in Infants Undergoing Cardiopulmonary Bypass. Pediatr Cardiol. 2022 Oct;43(7):1444-1454. doi: 10.1007/s00246-022-02866-4. Epub 2022 Mar 19. PMID 35305111
- See also: Nicklaus Children's Hospital — https://www.nicklauschildrens.org/home

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RiaSTAP | Saline
Started | 15 (First subject enrolled on 6-1-17.) | 15 (First subject enrolled on 6-1-17.)
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline is 15 in RiaSTAP and 15 in Saline solution.
Groups:
- Total: Total of all reporting groups
Arm/Group | RiaSTAP | Saline | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Mixed Race | 2 | 0 | 2
  Race: Black/African American | 3 | 2 | 5
  Race: White | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Blood Loss After Surgery (Estimated Blood Loss (EBL))
Description: Primary outcome efficacy: Estimated blood loss (EBL); median; A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Thereafter, as per routine care, ROTEM analysis was performed at least every 30 minutes while in the OR, or sooner, at the discretion of the OR team. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algorithm.
Time Frame: Within 24 hours of surgery
Measure: Median (Inter-Quartile Range); unit: cc/kg
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
cc/kg | 35 [21 to 61] | 33 [26 to 48]

2. Primary Outcome: Post-operative 2 hr Hemoglobin (Hg) mg/dL Measure
Description: Post-operative 2 hr hemoglobin (Hg) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Thereafter, as per routine care, ROTEM analysis was performed at least every 30 minutes while in the OR, or sooner, at the discretion of the OR team. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algorithm.
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
mg/dL | 13.6 [11.0 to 15.2] | 12.5 [11.7 to 13.3]

3. Primary Outcome: Post-operative 24-hr Hemoglobin (Hg) mg/dL
Description: Post-operative 24-hr hemoglobin (Hg) between treatment and placebo. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Thereafter, as per routine care, ROTEM analysis was performed at least every 30 minutes while in the OR, or sooner, at the discretion of the OR team. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algorithm.
Time Frame: 24 hr
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
mg/dL | 13.8 [11.7 to 15.8] | 12.4 [11.0 to 14.7]

4. Primary Outcome: Post-operative 2 hr Hematocrit (HCT) Measure
Description: Post-operative 2 hr Hematocrit (HCT) between the treatment and placebo group.
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: percent of hematocrit
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
percent of hematocrit | 40.9 [32.7 to 43.5] | 35.9 [35.4 to 38.8]

5. Primary Outcome: Post-operative 24 hr Hematocrit (HCT) Measure
Description: Post-operative 24 hr Hematocrit (HCT) between the treatment and placebo group
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
percent | 38.9 [34.1 to 45.3] | 35.4 [32.9 to 42.8]

6. Primary Outcome: Post-operative 2 hr Platelets Count Test (PLT) 10K/uL
Description: Post-operative 2 hr Platelets Count Test (PLT) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algor
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: 10x10^3 platelets/uL
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
10x10^3 platelets/uL | 282.0 [234.0 to 309.0] | 224.0 [192.0 to 311.0]

7. Primary Outcome: Post-operative 24 hr Platelets Count Test (PLT) 10K/uL
Description: Post-operative 24 hr Platelets Count Test (PLT) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algo
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: 10x10^3 platelets/uL
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
10x10^3 platelets/uL | 249.0 [197.0 to 297.0] | 247.0 [189.0 to 300.0]

8. Primary Outcome: Post-operative 2 hr Prothrombin (PT) Seconds
Description: Post-operative 2 hr Prothrombin (PT) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Thereafter, as per routine care, ROTEM analysis was performed at least every 30 minutes while in the OR, or sooner, at the discretion of the OR team. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algorithm.
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
seconds | 17.0 [16.7 to 18.5] | 16.5 [15.8 to 17.2]

9. Primary Outcome: Post-operative 24 hr Prothrombin (PT) Seconds
Description: Post-operative 24 hr Prothrombin (PT) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Thereafter, as per routine care, ROTEM analysis was performed at least every 30 minutes while in the OR, or sooner, at the discretion of the OR team. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algorithm.
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
seconds | 16.0 [15.4 to 18.2] | 16.1 [14.9 to 17.1]

10. Primary Outcome: Post-operative 2 hr International Normalize Ratio (INR)
Description: Post-operative 2 hr International Normalize Ratio (INR) between the treatment and placebo group
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
ratio | 1.4 [1.3 to 1.5] | 1.4 [1.2 to 1.4]

11. Primary Outcome: Post-operative 24 hr International Normalize Ratio (INR)
Description: Post-operative 24 hr International Normalize Ratio (INR) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM ana
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
ratio | 1.3 [1.2 to 1.5] | 1.3 [1.2 to 1.4]

12. Primary Outcome: Post-operative 2 hr Partial Thromboplastin Time (PTT) Seconds
Description: Post-operative 2 hr Partial Thromboplastin Time (PTT) between the treatment and placebo group
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
seconds | 36.7 [33.7 to 41.1] | 35.2 [32.1 to 36.6]

13. Primary Outcome: Post-operative 24 hr Partial Thromboplastin Time (PTT) Seconds
Description: Post-operative 24 hr Partial Thromboplastin Time (PTT) between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analys
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
seconds | 35.5 [34.1 to 38.6] | 31.5 [30.3 to 35.5]

14. Primary Outcome: Post-operative 2 hr Fibrinogen mg/dL
Description: Post-operative 2 hr Fibrinogen between the treatment and placebo group. A transfusion algorithm was developed based on three previous studies, modified for pediatrics. Clinically significant bleeding requiring treatment was defined as a rate >10 cc kg-1 hr-1 calculated every 15 minutes while in the OR, measured by blood in the suction canister. In cases of continued bleeding following randomization to HFC or placebo, cryoprecipitate was considered for fibrinogen <200 mg/dL or FIBTEM MCF <7 mm. Thereafter, as per routine care, ROTEM analysis was performed at least every 30 minutes while in the OR, or sooner, at the discretion of the OR team. Once the patient left the OR, ROTEM was performed at least every 60 minutes for the first 6 hours or until clinically significant bleeding had stopped. Blood products transfused after CPB separation were based on a pre-defined protocol. Recommended volumes of each therapy were based on pre-defined formulae and a ROTEM analysis algorithm.
Time Frame: 2 hour
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
mg/dL | 258.0 [238.0 to 338.0] | 330.0 [281.0 to 385.0]

15. Primary Outcome: Post-operative 24 hr Fibrinogen mg/dL
Description: Post-operative 24 hr Fibrinogen between the treatment and placebo group
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
mg/dL | 416.5 [318.5 to 512.0] | 403.0 [324.0 to 465.0]

16. Secondary Outcome: Post-Operative Respiratory Failure Adverse Events
Description: Patients who suffered from respiratory failure post operatively.
Time Frame: 24 hours after surgery
Measure: Number; unit: participants
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
participants | 3 | 3

17. Secondary Outcome: Post-operative Thrombus Adverse Events
Description: Patient who suffered from Thrombus events post-operatively.
Time Frame: within 24 hours of surgery
Measure: Number; unit: participants
Arm/Group | RiaSTAP | Saline
Number analyzed (Participants) | 15 | 15
participants | 4 | 2

ADVERSE EVENTS:
Time Frame: 24 hours after surgery;
Description: There were no other adverse events measured
Groups:
- RiaStap: RiaStap_Treatment received an infusion of RiaSTAP, right after the termination of CPB at a dose of 70 mg/kg.
- Placebo: Placebo_Treatment received a placebo of Normal Saline 0.9% (NS) during the same time period. The volume of NS was calculated to be the same volume that would be used IF the patient were receiving RiaSTAP.
Arm/Group | RiaStap | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 7/15 | 5/15
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RiaStap (N=15) | Placebo (N=15)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Thrombus (Cardiac disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT02822599/Prot_SAP_000.pdf